CLINICAL TRIAL: NCT04878458
Title: Effectiveness and Safety of Phacotrabeculectomy and Phacogoniotomy in Advanced Primary Angle-closure Glaucoma: a Multicenter Randomized Controlled Trial
Brief Title: Phacotrabeculectomy Versus Phacogoniotomy (PVP) in Advanced Primary Angle-closure Glaucoma
Acronym: PVP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: The Second Affiliated Hospital of Harbin Medical University (Other); West China Hospital (Other); First Hospital of Shijiazhuang City (Other); Union hospital of Fujian Medical University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Handan City Eye Hospital (Unknown); Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Director of Clinical Research Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021KYPJ090
Record Dates: First submitted 2021-05-06; First posted 2021-05-07 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma, Angle-Closure
Keywords: Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Phacoemulsification; Trabeculectomy

STUDY DESIGN:
Intervention Model Description: multicenter, parallel, open, non-inferior randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEI+GSL+GT (Experimental): Sixty-two patients with advanced primary angle-closure glaucoma will receive phacoemulsification with intraocular lens implantation combined with goniosynechialysis and goniotomy.
  Interventions: Procedure: phacoemulsification with intraocular lens implantation combined with goniosynechialysis and goniotomy
- PEI+Trab (Experimental): Sixty-two patients with advanced primary angle-closure glaucoma will receive phacoemulsification with intraocular lens implantation combined with trabeculectomy.
  Interventions: Procedure: phacoemulsification with intraocular lens implantation combined with trabeculectomy

INTERVENTIONS:
Procedure: phacoemulsification with intraocular lens implantation combined with goniosynechialysis and goniotomy — The patients enrolled underwent phacoemulsification with intraocular lens implantation combined with goniosynechialysis and goniotomy.
  Arms: PEI+GSL+GT
Procedure: phacoemulsification with intraocular lens implantation combined with trabeculectomy — The patients enrolled underwent phacoemulsification with intraocular lens implantation combined with trabeculectomy.
  Arms: PEI+Trab

SUMMARY:
A multicenter, parallel, open, non-inferior randomized controlled trial was conducted to compare the effectiveness and safety of phacotrabeculectomy and phacogoniotomy in the treatment of advanced primary angle closure glaucoma, so as to provide a better surgical alternative.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide, and primary angle closure glaucoma (PACG) accounted for the majority particularly in Asia and China. The preferred treatment method is anti-glaucoma surgery-trabeculectomy (Trab) combined with lens extraction. Phacotrabeculectomy has become the first-line choice of anti-glaucoma suregery in the treatment of advanced PACG. However, it was not an ideal method due to the bleb-related complications and troublesome postoperative nursing, as well as the difficulty for surgeons, caused by trabeculectomy. However, recent studies revealed that the phacoemulsification with intraocular lens implantation (PEI) combined with goniosynechialysis (GSL) has achieved efficacy in the treatment of PACG.

With the advent of minimally invasive glaucoma surgeries (MIGS), there is an increasing number studies indicating the MIGS performed great efficacy in the treatment of primary open angle glaucoma. While,there were a few small-sampled retrospective studies which showed therapeutic effects in PACG. The GSL plus goniotomy (GT) could achieve great efficacy in lowering the intraocular pressure of PACG patients. However, there is still a lack of high quality and high-level randomized controlled trials.

Therefore, this study intends to conduct a multicenter, parallel, open, non-inferior randomized controlled trial to compare the effectiveness and safety of PEI+ Trab and PEI+GSL+GT in the treatment of advanced PACG, so as to provide a better surgical treatment for PACG.

ELIGIBILITY:
* Inclusion criteria

  1. Aged 40-80 years;
  2. Diagnosed with advanced PACG: meet with (1) (2) (3) or (1) (2) (4)

     1. At least 180-degree PAS under gonioscopy and it should cover the nasal and inferior quadrants for surgical purposes;
     2. IOP >21 mmHg with or without anti-glaucoma medication;
     3. Obvious glaucomatous optic neuropathy (cup-to-disc [C/D] ratio≥0.7, or C/D asymmetry > 0.2, or the rim width at the superior and inferior temporal < 0.1 vertical diameters of optic disc);
     4. With glaucomatous visual field defects, such as nasal step, arcuate scotoma, and paracentral scotoma on a reliable Humphrey analyzer using SITA-Standard 24-2 or 30-2 algorithm; mean deviation ≤ -12dB;
  3. Clinically obvious cataract and uncorrected visual acuity (UCVA) <0.63 (Early Treatment Diabetic Retinopathy Study, [ETDRS] chart), or need lens extraction assessed by a clinician;
  4. Voluntarily participate in study and provide signed informed consent.
* Exclusion criteria a. History of ocular surgery (other than laser iridotomy or laser iriplasty) or trauma; b. With other types of glaucoma; (i.e. open angle glaucoma, secondary angle-closure glaucoma, steroidal glaucoma, angle regression glaucoma, neovascular glaucoma, nanophthalmos, pseudoexfoliation syndrome) c. The International Standardized Ratio > 3.0 for patients receiving warfarin or anticoagulant therapy before surgery; d. With retinal disease that affects the collection of ocular parameters; f. Monophthalmia (best-corrected visual acuity [BCVA] <0.01 in the non-study eye); g. With other serious systemic diseases; h. Pregnant or lactating women * If both eyes are eligible for the study, the eye with the worse UCVA will be recruited.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean change of intraocular pressure | Postoperative 12, 24, 36 months.
  Change from baseline IOP after surgery using Goldmann or non-contact tonometer.

SECONDARY OUTCOMES:
Cumulative success rate of surgery | 12, 24, 36 months
  (i) Complete success is defined as the postoperative IOP between 5 and 18 mmHg, and 20% reduction from baseline with no need for IOP-lowering medication.
  (ii) Qualified success is defined as the postoperative IOP between 5 and 18 mmHg, and 20% reduction from baseline with or without IOP-lowering medication.
Intraoperative and postoperative complications | 0, 1, 7 day. 1, 3, 6, 12, 18, 24, 30, 36 months
  For example, shallow anterior chamber, hyphema, persistent hypotony, corneal endothelium decompensation, endophthalmitis, and other filtering bleb-related complications.
Anti-glaucomatous medications | 0, 1, 7 day. 1, 3, 6, 12, 18, 24, 30, 36 months
  Numbers and types of anti-glaucomatous medications

OTHER OUTCOMES:
Visual acuity | 0, 1, 7 day. 1, 3, 6, 12, 18, 24, 30, 36 months
  Uncorrected and best corrected visual acuity will be documented using ETDRS chart.
Degree of peripheral anterior synechia | 3, 12, 24, 36 months
  The peripheral anterior synechia is checked using gonioscopy.
Corneal endothelial cell counting | 0, 12, 24, 36 months
  Corneal endothelial cell counting will be documented using specular microscope.
Visual field | 0, 12, 24, 36 months
  Visual field examination is performed using Humphrey analyzer.
Optic nerve head morphology and retinal parameters | 0, 12, 24, 36 months
  Optic nerve head morphology and retinal parameters based on optical coherence tomography (Cirrus 5000, Zeiss, CA, USA or Spectralis, Heidelberg, Germany)
Measurement of quality of life | 0, 12, 24, 36 months
  Quality of life is measured with EQ-5D-5L questionnaire.
Filtering bleb classification | 12, 24, 36 months
  Filtering bleb classification based on Indiana Bleb Appearance Grading Scale
Time-consuming of operation and the surgery cost | 1 day
  Time-consuming of operation and the surgery cost are based on the electronic healthy system.

CONTACTS AND LOCATIONS:
Overall Officials: Xiulan Zhang, MD, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (2):
- China (2):
  - Zhongshan Ophthalmic Center, Guangzhou, Guangdong
  - Zhongshan Ophthalmic Center, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Husain R, Do T, Lai J, Kitnarong N, Nongpiur ME, Perera SA, Ho CL, Lim SK, Aung T. Efficacy of Phacoemulsification Alone vs Phacoemulsification With Goniosynechialysis in Patients With Primary Angle-Closure Disease: A Randomized Clinical Trial. JAMA Ophthalmol. 2019 Oct 1;137(10):1107-1113. doi: 10.1001/jamaophthalmol.2019.2493. PMID 31294768
- [Background] Barry M, Alahmadi MW, Alahmadi M, AlMuzaini A, AlMohammadi M. The Safety of the Kahook Dual Blade in the Surgical Treatment of Glaucoma. Cureus. 2020 Jan 16;12(1):e6682. doi: 10.7759/cureus.6682. PMID 31976190
- [Background] Tanito M, Sugihara K, Tsutsui A, Hara K, Manabe K, Matsuoka Y. Midterm Results of Microhook ab Interno Trabeculotomy in Initial 560 Eyes with Glaucoma. J Clin Med. 2021 Feb 17;10(4):814. doi: 10.3390/jcm10040814. PMID 33671386
- [Background] Grover DS, Smith O, Fellman RL, Godfrey DG, Gupta A, Montes de Oca I, Feuer WJ. Gonioscopy-assisted Transluminal Trabeculotomy: An Ab Interno Circumferential Trabeculotomy: 24 Months Follow-up. J Glaucoma. 2018 May;27(5):393-401. doi: 10.1097/IJG.0000000000000956. PMID 29613978
- [Background] Dorairaj S, Tam MD, Balasubramani GK. Two-Year Clinical Outcomes of Combined Phacoemulsification, Goniosynechialysis, and Excisional Goniotomy For Angle-Closure Glaucoma. Asia Pac J Ophthalmol (Phila). 2020 Oct 6;10(2):183-187. doi: 10.1097/APO.0000000000000321. PMID 33031110
- [Background] Tham CC, Kwong YY, Baig N, Leung DY, Li FC, Lam DS. Phacoemulsification versus trabeculectomy in medically uncontrolled chronic angle-closure glaucoma without cataract. Ophthalmology. 2013 Jan;120(1):62-7. doi: 10.1016/j.ophtha.2012.07.021. Epub 2012 Sep 15. PMID 22986111
- [Result] Song Y, Li F, Zhang X. Response: Comment on "Phacogoniotomy versus phacotrabeculectomy for advanced primary angle-closure glaucoma with cataract: A randomized non-inferiority trial". Asia Pac J Ophthalmol (Phila). 2024 May-Jun;13(3):100076. doi: 10.1016/j.apjo.2024.100076. Epub 2024 May 23. No abstract available. PMID 38795868
- [Result] Song Y, Lin F, Lv A, Zhang Y, Lu L, Xie L, Tang G, Yuan H, Yang Y, Xu J, Lu P, Xiao M, Zhu X, Yan X, Song W, Li X, Zhang H, Li F, Wang Z, Jin L, Gao X, Liang X, Zhou M, Zhao X, Zhang Y, Chen W, Wang N, Tham CC, Barton K, Park KH, Aung T, Weinreb RN, Tang L, Fan S, Lam DSC, Zhang X; PVP Study group. Phacogoniotomy versus phacotrabeculectomy for advanced primary angle-closure glaucoma with cataract: A randomized non-inferiority trial. Asia Pac J Ophthalmol (Phila). 2024 Jan-Feb;13(1):100033. doi: 10.1016/j.apjo.2023.100033. Epub 2023 Dec 26. PMID 38383075
- [Derived] Song Y, Fan S, Tang L, Lin F, Li F, Lv A, Li X, Wen T, Lu L, Xiao M, Xie L, Zhu X, Tang G, Zhang H, Yan X, Yuan H, Song W, Yang Y, Xu J, Zhou F, Wang Z, Jin L, Liang X, Zhou M, Zhao X, Chen W, Park KH, Barton K, Aung T, Tham CC, Lam DSC, Weinreb RN, Wang N, Zhang X; PVP Study Group. Two-Year Outcomes of Phacogoniotomy vs Phacotrabeculectomy for Advanced Primary Angle-Closure Glaucoma With Cataract: A Noninferiority Randomized Clinical Trial. JAMA Ophthalmol. 2025 Jun 1;143(6):462-469. doi: 10.1001/jamaophthalmol.2025.0685. PMID 40244620
- [Derived] Song Y, Song W, Zhang Y, Zhang H, Xiao M, Zhao X, Lv A, Yan X, Lu P, Zhu X, Gao X, Hu K, Zhang Y, Liang X, Zhang X, Tang G, Lu L, Zhou M, Fan S, Xie L, Jin L, Tang L, Yuan H, Zhang X; PVP Study group. Efficacy and safety of phacotrabeculectomy versus phacogoniotomy in advanced primary angle-closure glaucoma: study protocol for a multicentre non-inferiority randomised controlled trial (PVP Study). BMJ Open. 2021 Dec 8;11(12):e056876. doi: 10.1136/bmjopen-2021-056876. PMID 34880029